CLINICAL TRIAL: NCT00643942
Title: Staining in a Healthy, Non-Dry Eye Population
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Judy Vittitoe, Alcon
Other Study IDs: C-06-23
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2008-03

CONDITIONS: Normal Healthy Eyes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: No intervention required

INTERVENTIONS:
Other: No intervention required

SUMMARY:
The clinical objective of this study is to quantify the levels of corneal and conjunctival staining in a healthy, non-dry eye population. This is a descriptive study without test article administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy eyes

Exclusion Criteria:

* Age related

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with normal healthy eyes
Sampling Method: Probability Sample
Enrollment: 120
Dates: Start 2007-06; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Corneal fluorescein staining scores

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio, San Antonio, Texas, United States